CLINICAL TRIAL: NCT03557866
Title: Kinematic Parameters of Running in Individuals With Pronated Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, principal investigator, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 380/17
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pronation; Ankle
Keywords: foot posture; running; foot index
MeSH Terms: interventions — Running

STUDY DESIGN:
Intervention Model Description: two groups. Individuals with and without pronated foot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pronated group (Experimental): individuals with pronated foot
  Interventions: Diagnostic Test: running
- control group (Active Comparator): individuals with normal foot posture
  Interventions: Diagnostic Test: running

INTERVENTIONS:
Diagnostic Test: running — individuals will be asked to run for 5 km in self selected speed
  Other Names: kinematic parameters of running

SUMMARY:
The aim of the study is to examine the kinematic parameters of individuals with pronated foot compared with individuals with normal foot

DETAILED DESCRIPTION:
Individual with and without pronated foot will be recruited. Pronation will be defined according to navicular drop test. Inclusion criteria : individual who run on a regular basis at least 3 times per week for one hour, can run 5 Km in less then 40 minutes, without past injuries during the last year of Achilles tendon or other lower extremities pain.

Individuals will be asked to run for 5 Km in self selected velocity. The Milestone pod device will be used to monitor kinematic parameters.

functional test will be conducted before and after the running as follows: heel raise test and one leg hop for distance test.

ELIGIBILITY:
Inclusion Criteria:

* running on a daily basis at least 3 times per week with minimum of 1 hour
* capable to run 5 km in less then 40 minutes
* willing to participate in the study

Exclusion Criteria:

* previous surgery in lower extremities
* Achilles tendon pain during the last year

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
stride length | up to 6 months
  stride length in cm
cadence | up to 6 months
  steps per minute

SECONDARY OUTCOMES:
velocity | up to 6 months
  running velocity in Km/hour
heel raise test | up to 6 months
  how many good heel raise till fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PHd, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
the results of the study will be analysed. a paper will be submitted to international journal with study description including methods, examination protocol and results
Supporting Information: Study Protocol, CSR
Time Frame: following completion of data collection
Access Criteria: according to journal policy

REFERENCES:
- [Result] McPoil TG, Cornwall MW, Medoff L, Vicenzino B, Fosberg KK, Hilz D. Arch height change during sit-to-stand: an alternative for the navicular drop test. J Foot Ankle Res. 2009 May 18;2:17. doi: 10.1186/1757-1146-2-17. PMID 19450247
- [Result] Murley GS, Menz HB, Landorf KB. Foot posture influences the electromyographic activity of selected lower limb muscles during gait. J Foot Ankle Res. 2009 Nov 26;2:35. doi: 10.1186/1757-1146-2-35. PMID 19939283